CLINICAL TRIAL: NCT05252832
Title: Evaluation of the Efficacy of the Superficial Cervical Plexus Block in Reducing Pain Associated With Internal Jugular Central Lines
Brief Title: Superficial Cervical Plexus Block for IJCL Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cleveland Clinic Akron General (Other)
Responsible Party: Principal Investigator, Robert Stenberg, Principle Investigator, Ultrasound Director, Assistant Professor, Emergency Medicine Physician, Cleveland Clinic Akron General
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21003
Record Dates: First submitted 2021-12-07; First posted 2022-02-23 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Superficial Cervical Plexus Block; Pain
Keywords: Superficial Cervical Plexus Block; Pain Management
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: Participant blinded block randomization of the control local infitrate (Arm 1) and the experimental SCPB (Arm 2).
Who Masked: Participant
Masking Description: Participants will be masked to the anesthesia route selected until after they report their pain scale report. Care provider cannot be blinded in order to complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Local Infitrate (Active Comparator)
  Interventions: Procedure: Local Infiltrate
- SCPB (Experimental)
  Interventions: Procedure: Superficial Cervical Plexus Block

INTERVENTIONS:
Procedure: Superficial Cervical Plexus Block — Location of injection for block.
  Arms: SCPB
Procedure: Local Infiltrate — Local infiltration location.
  Arms: Local Infitrate

SUMMARY:
This is a prospective randomized trial evaluating the effect of SCPB on reported patient pain following IJCL placement as compared to local infiltrate.

DETAILED DESCRIPTION:
The goal of this study is to determine if SCPBs provide more pain control than local infiltrate of anesthetic for internal jugular venous cannulation. The investigators hypothesis that patients who receive the SCPB will have a lower VAS rating on average than those who receive local infiltration following internal jugular venous cannulation. To test this, the investigators will be approaching eligible patients for inclusion in a research study. If the patients consent, the patients will be randomly assigned the standard of care treatment or the SCPB. The investigators will then ask the patients to rate pain following insertion of the central line. The investigators will also evaluate different aspects of the patient's hospital course to evaluate their outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 years and older, and;
* Present to the Akron General Emergency Department (Main) between March 1, 2021 and December 1, 2022, and;
* Require IJVC as a part of their clinical care.

Exclusion Criteria:

* Patients who are intubated; or
* Patients who undergo CPR; or
* Patients who have an allergy to lidocaine or bupivacaine; or
* Patients who have a contraindication to receiving a superficial cervical plexus block such as cellulitis over Erb's point or the internal jugular vein, abnormal anatomy, or prior surgery to the area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale Rating | 30 minutes post central line placement
  The average Visual Analog Scale (VAS) rating in patients who receive the SCPB during internal jugular venous cannulation versus the average VAS in patients receiving local infiltration. The scale is from 0-10, with 0 meaning no pain and 10 meaning the most pain I have ever experienced.

SECONDARY OUTCOMES:
Complications | Duration of emergency department and inpatient encounter, typically no more than 7 days.
  To determine if SCPBs are associated with higher complication rates than local infiltration with internal jugular venous cannulation. Complications will be defined as arterial injury, lacerations of the vena cava, mediastinal vessels, and right atrium, hematoma formation, retained guide wire, pulmonary complications including pneumothorax, pneumomediastinum, chylothorax, tracheal injury, injury to the recurrent laryngeal nerve, and air embolus, tracheal injury, arrhythmia, cardiac arrest, device dysfunction, device infection, and venous thrombosis.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Stenberg, MD, Principal Investigator — Cleveland Clinic Akron General
Locations (1):
- Cleveland Clinic Akron General, Akron, Ohio, United States

IPD SHARING:
Plan to Share IPD: No